CLINICAL TRIAL: NCT03973788
Title: Immediate and Short-term Effects of Single-session Repetitive Transcranial Magnetic Stimulation on Pain Thresholds In Patients With Chronic Low Back Pain - A Pilot Study
Brief Title: Effects of Repetitive Transcranial Magnetic Stimulation on Pain Thresholds in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Sharon Wang-Price, Professor, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20394
Record Dates: First submitted 2019-05-30; First posted 2019-06-04 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low Back Pain (CLBP)
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Pre and post test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): repetitive transcranial magnetic stimulation
  Interventions: Procedure: repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Procedure: repetitive transcranial magnetic stimulation (rTMS) — A single section of rTMS (2,000 pulses)

SUMMARY:
Chronic low back pain (CLBP) is a common reason for which patients are treated with opioids. Because the misuse of prescription opioids has become a serious problem in the Uinted States, finding effective alternative non-pharmaceutical interventions for chronic pain management has become an urgent matter. A phenomenon termed central sensitization (i.e. mal-adaption of the brain) has been hypothesized to be an underlying mechanism for the development of chronic pain, leading to sensory hypersensitivity to extremal stimuli. Therefore, non-invasive brain stimulation, such as repetitive transcranial magnetic stimulation (rTMS) may be an effective intervention to regulate brain excitability, thus reducing chronic pain. However, research has shown inconclusive evidence regarding the rTMS effects on chronic pain reduction, partly due to the heterogeneity of participants in studies to date. Therefore, the primary purpose of this study is to investigate the immediate and short-term effects of rTMS on neurosensory changes (i.e., pain thresholds) in patients with CLBP. The secondary purpuse of the study is to explore the relationship between changes of cortical excitability (TMS parameters) and changes of pain thresholds after the rTMS intervention in patients with CLBP.

DETAILED DESCRIPTION:
Research Design

A pre- and post-test research design will be used to examine the immediate and one-week carry-over effects of a single-session of rTMS intervention on individuals with CLBP. The primary outcome measures, including PPT, cold pain threshold (CPT), heat pain threshold (HPT), and heat-generated temporal summation (TS), will be collected three times: before the rTMS intervention, immediately after the intervention, and one week after the intervention.

Participants

Eligible participants are adults 18 years of age or older and who have had LBP for more than 6 months. According to the Centers for Disease Control and Prevention, chronic pain is defined as pain lasts more than 3 months or past the time of normal tissue healing. In order to ensure the development of central sensitization in the investigator's participants, only individuals with LBP for more than 6 months will be enrolled in this study.

Participants will be excluded from the study if they have previous low back surgery, systemic joint disease (e.g. rheumatoid arthritis), evidence of red flags (e.g. fracture, infection, tumor, cauda equina syndrome), cancer, neurological disorders, neuropathy, Raynaud's Disease or pregnancy, and inability to maintain the testing and treatment positions (i.e. sitting, supine hook-lying and prone-lying) for 15 minutes at a time. Additional exclusion criteria for the rTMS intervention include: 1) history of significant head trauma, 2) electrical, magnetic, or mechanical implantation (e.g. cardiac pacemakers or intracerebral vascular clip), 3) metal implantation in the head and neck areas, 4) history of seizures or unexplained loss of consciousness, 5) immediate family member with epilepsy, 6) use of seizure threshold lowering medicine, 7) current abuse of alcohol or drugs, and 8) history of psychiatric illness requiring medication controls.

Procedure

After the participant is enrolled the study, the participant will be asked to complete an intake form, collecting their demographic data (age, gender, height, weight, occupation, hand dominance), past medical history, and questions related to their low back pain (onset, injury mechanism if any, location, duration, type, and nature). In addition, 4 self-reported questionnaires will be collected from all of the participants before the rTMS treatment, including pain intensity determined using the NPRS, disability determined using the Modified Oswestry Low Back Pain Disability Questionnaire quality of life determined by the Patient-Reported Outcomes Measurement Information System® - short form (PROMIS-29), and severity of central sensitization determined by the Central Sensitization Inventory (CSI ). These questionnaires are commonly used in research studies of chronic pain or CLBP.

1. Pain Threshold Tests:

   All participants will undergo a battery of tests to determine their sensory thresholds, including pressure, cold and heat pain thresholds and heat-generated temporal summation (TS). The pain thresholds and TS will be measured from three sites: the most painful point of low back, as well as the web space (WS) and the tibialis anterior (TA) of the painful side. Those who report no pain difference between the right and left low back, pain thresholds will be measured from the right side. The TA testing site will be in the muscle belly of the TA, approximately 2.5 cm lateral and 5 cm inferior to the tibial tubercle. The WS and TA sites were chosen because they are the most commonly selected sites in research studies for chronic pain. In addition, the first interosseous index (FDI) is located in the WS, where is the target site for the TMS assessment and intervention.

   Pressure pain threshold (PPT) testing: A hand-held computerized pressure algometer (Medoc ltd., Ramat Yishai, Israel) will be used to measure the PPTs. The algometer consists of a 1-sqaure centermeter round tip which will be pressed vertically on the target location of the muscle. To provoke the patient's pain or discomfort, pressure will be increased at a rate of 40 kPa/sec until the participant feels pain as indicated by pressing a patient safety unit. The limit of pressure threshold will be set at 800 kPa, meaning that a pressure exceeding 800 kPa will be cut off to minimize tissue damage. If the participant does not push the button at 800 kPa, a value of 800 is used as the threshold value. Three trials of PPT testing will be administered to each testing site, and the average of the three trials will be used for data analysis.

   Cold and heat pain threshold testing: A Medoc TSA II Neurosensory Analyzer (Medoc ltd., Ramat Yishai, Israel) will be used to measure heat and cold pain thresholds. All thermal pain threshold tests will be obtained with ramped stimuli (0°5 C/s) which can be terminated when the participant presses a safety button. Cut-off temperatures will be set 0 and 52°C, and the baseline temperature will be set at 32°C (i.e., average skin temperature). The contact area of the thermode is 23mmx30mm. All thermal pain threshold tests will be demonstrated first at an area somewhere other than the three testing sites. Three trials of thermal pain threshold tests will be administered per testing site and the average of the three trials will be used for statistical analysis.

   Heat-generated temporal summation (TS) testing: The instrument used for measuring cold and heat pain thresholds will be used for the heat-generated TS test. During TS testing, 10 consecutive heat pulses of 0.5 sec duration will be delivered at an inter-stimulus interval of 2.5 sec. The temperature of the heat stimuli will increase from 40°C as a baseline temperature and inter-stimulus temperature, to 48°C at a rate of 8°C/sec. Participants will be asked to rate their pain intensity of each heat pulse on the NPRS of 0-100 (0 being no pain, 100 being unbearable pain). The TS score will be calculated by averaging the pain rating for the 10th stimulus and the 5th stimulus minus the 1st pain rating, with higher score indicating greater hypersensitivity of pain.
2. Cortical Excitability Assessment

   A series of single pulse generated from a TMS machine (Rapid2, Magstim Co., UK) will be used to determine corticospinal excitability. Because the rTMS intervention will target the M1 area, specifically in the area corresponding to the FDI muscle, motor evoked potentials (MEPs), namely electromyographic (EMG) activity, will be recorded from the FDI muscle to determine the "hot spot" for the rTMS intervention. A hot spot is defined as the site at which the largest MEP amplitude is obtained at the lowest TMS stimulation intensity.

   First, a pair of surface EMG electrodes will be placed on the FDI muscle when the participant is seated on a reclining chair and wearing a pair of earplugs to reduce their awareness of noise from the rTMS equipment. Similar to the pain threshold testing on the low back, EMG activity will be measured from FDI muscle on the same side of the patient as the LBP. For those who report no difference in LBP between sides, EMG data will be recorded from the FDI of the right hand. The Mega 600 EMG machine (Mega Electronics Ltd., Finland) will be used to collect EMG data at a sampling rate of 2,000Hz and bandpass-filtered at 15-500Hz. During the cortical excitability assessment, each participant will wear a Lycra swimming cap with a pre-marked grid. The intensity of TMS will begin at 40% of maximum stimulator output and then will be increased gradually to yield a MEP from the FDI until a 'hot spot' is observed. Next, the resting motor threshold (RMT) will be defined. RMT is the stimulation intensity which yields a peak-to-peak amplitude of MEP larger than 50 μV in 5 out of 10 consecutive trials. Once the RMT is determined, the stimulation intensity will be set at 120% of RMT and 10 stimulations will be delivered to the hot-spot. The 10 supra-threshold MEP amplitudes recorded from the FDI will be averaged and the average will be used for the representation of corticospinal excitability.
3. rTMS Intervention

After the corticospinal excitability assessment, participants will receive 10Hz rTMS delivered to the hot-spot contralateral to the painful side in the form of twenty 10-second pulse trains (a total of 2,000 pulses) with a 50-second inter-train interval. The rTMS will be delivered via an air-filled coil (see figure to the right). The stimulation intensity will be set at 90% of RMT. After the rTMS intervention, the participant's corticospinal excitability will be re-assessed using the single-pulse TMS method as described earlier.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Have LBP for more than 6 months

Exclusion Criteria:

* Previous low back surgery, systemic joint disease (e.g. rheumatoid arthritis),
* Fracture,
* Infection
* Tumor or cancer
* Cauda equina syndrome
* neurological disorders
* Neuropathy
* Raynaud's Disease
* pregnancy,
* Inability to maintain the testing and treatment positions (i.e. sitting, supine hook-lying and prone-lying) for 15 minutes at a time.
* History of significant head trauma,
* Electrical, magnetic, or mechanical implantation (e.g. cardiac pacemakers or intracerebral vascular clip)
* Metal implantation in the head and neck areas
* History of seizures or unexplained loss of consciousness,
* Immediate family member with epilepsy
* Use of seizure threshold lowering medicine
* Current abuse of alcohol or drugs
* History of psychiatric illness requiring medication controls

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Pain thresholds | before intervention, immediate after intervention, and one week after intervention
  pressure pain thresholds, cold pain thresholds, and heat pain thresholds, and heat-generated temporal summation using a A Medoc TSA II Neurosensory Analyzer (Medoc ltd., Ramat Yishai, Israel).

SECONDARY OUTCOMES:
Cortical Excitability | before intervention and immediate after intervention
  10 supra-threshold motor evoked potentials (MEP) amplitudes recorded from the first interosseous index (FDI) muscle using a transcranial magnetic stimulation machine (Rapid2, Magstim Co., UK)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Wang-Price, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the corresponding author, Sharon Wang-Price. The data are not publicly available due to their containing information that could compromise the privacy of research participants.